CLINICAL TRIAL: NCT03355196
Title: A Randomized, Placebo Controlled, Subject and Investigator Blinded, first-in- Human, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics After Intra-articular Injection of LRX712 Into the Knee of Osteoarthritic Patients
Brief Title: First-in-human, Safety, Tolerability and Pharmacokinetics Study of LRX712 in Osteoarthritic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLRX712X2101
Record Dates: First submitted 2017-11-17; First posted 2017-11-28 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-05

CONDITIONS: Patients With Moderate Knee Osteoarthritis (30 - 65 Years)
Keywords: Osteoarthritic patients; Cartilage; Safety

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LRX712 (Experimental): LRX712 given intra-articularly
  Interventions: Drug: LRX712
- Placebo (Placebo Comparator): Placebo given intra-articularly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LRX712 — Ascending single dose on Day 1
  Arms: LRX712
Drug: Placebo — Ascending single dose on Day 1
  Arms: Placebo

SUMMARY:
This study is designed to evaluate, for the first time in humans, safety and tolerability of single ascending doses of intra-articular (i.a.) injections of LRX712 into the knee of patients with moderate osteoarthritis (OA), in order to support the further clinical development. This study will also allow establishment of the systemic and local pharmacokinetics (PK) of LRX712 and the exploration of biomarkers of cartilage breakdown and regeneration in OA patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, 30 to 65 years of age inclusive, and in good health as determined by medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* At screening, and at baseline vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed in the sitting position after the subject has rested for at least three minutes, and again (when required) after three minutes in the standing position as outlined in the SOM.

Sitting vital signs should be guided by the following ranges:

* body temperature between 35.0-37.5 °C
* systolic blood pressure 90-139 mm Hg
* diastolic blood pressure 50-89 mm Hg
* pulse rate, 40 - 90 bpm • Subjects must weigh at least 50 kg to participate in the study, and must have a body mass index (BMI) within the range of 18 - 32 kg/m2. BMI = Body weight (kg) / [Height (m)]

Exclusion Criteria:

* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant.
* Pregnant or nursing (lactating) women
* Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days, whichever is longer; or longer if required by local regulations
* A history of clinically significant ECG abnormalities, or any of the following ECG abnormalities at screening and baseline

  * PR > 200 msec
  * QRS complex > 120 msec
  * QTcF > 450 msec (males)
  * QTcF > 460 msec (females)
* Known family history or known presence of long QT syndrome

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) of LRX712 after a single intra-articular (i.a.) injection in Osteoarthritic (OA) patients | Day 29
  To evaluate Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) of LRX712 after a single i.a. injection in osteoarthritic patients

SECONDARY OUTCOMES:
Time to Reach the Maximum Plasma Concentration (Tmax) | pre-dose to 29 days post-dose
  To evaluate LRX712 and metabolite MAE344 pharmacokinetics in plasma - Time to Reach the Maximum Plasma Concentration (Tmax)
Maximum Observed Plasma Concentration (Cmax) | pre-dose to 29 days post-dose
  To evaluate LRX712 and metabolite MAE344 pharmacokinetics in plasma - Maximum Observed Plasma Concentration (Cmax)
Area Under the Plasma Concentration-time Curve From 0 to the Last Measurable Concentration (AUClast) | pre-dose to 29 days post-dose
  To evaluate LRX712 and metabolite MAE344 pharmacokinetics in plasma - Area Under the Plasma Concentration-time Curve From 0 to the Last Measurable Concentration (AUClast)
Area under the plasma concentration-time curve from time zero to infinity (AUCinf) | pre-dose to 29 days post-dose
  To evaluate LRX712 and metabolite MAE344 pharmacokinetics in plasma - Area under the plasma concentration-time curve from time zero to infinity (AUCinf)
Half-life (T1/2) | pre-dose to 29 days post-dose
  To evaluate LRX712 and metabolite MAE344 pharmacokinetics in plasma - Half-life (T1/2)
CL/F - Total clearance | pre-dose to 29 days post-dose
  To evaluate LRX712 and metabolite MAE344 pharmacokinetics in plasma - CL/F - Total clearance
Vz/F - Volume of Distribution | pre-dose to 29 days post-dose
  To evaluate LRX712 and metabolite MAE344 pharmacokinetics in plasma - Vz/F - Volume of Distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CLRX712X2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17606
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=381